CLINICAL TRIAL: NCT05662878
Title: Evaluation of Hand Strength and Spasticity in Hemiplegic Patients Using Hand-Finger Robot Device
Brief Title: Evaluation of Hand Strength and Spasticity in Hemiplegic Patients
Status: Completed | Type: Observational
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Sevda Adar, Principal Investigator, Afyonkarahisar Health Sciences University
Other Study IDs: HemiHFR22
Record Dates: First submitted 2022-12-15; First posted 2022-12-23 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Neurological Rehabilitation; Stroke; Upper Extremity Problem
Keywords: Hemiplegia; Spasticity; Hand Grip Strength; Finger-Hand Robot
MeSH Terms: conditions — Stroke; Hemiplegia; Muscle Spasticity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient Group: Hemiplegic Patients
  Interventions: Other: Assessment of Hand Strength and Spasticity
- Control Group: Healthy Individuals
  Interventions: Other: Assessment of Hand Strength and Spasticity

INTERVENTIONS:
Other: Assessment of Hand Strength and Spasticity — Assessment of Hand Strength and Spasticity

SUMMARY:
The aim in this study is to evaluate spasticity and hand grip strength with a finger hand robot in the Turkish population.

DETAILED DESCRIPTION:
Spasticity has been defined as "irregular sensorimotor control resulting from upper motor neuron lesion manifesting as intermittent or sustained involuntary activation of muscles".

The commonly used tools in the evaluation of spasticity are subjective clinical scales, including Ashworth Scale (AS), Modified AS (MAS), Tardieu Scale (TS), Modified TS (MTS), and Tone Assessment Scale (TAS). Current scales are based on the clinician's perception of the patient assessing spasticity through their perceptions, experience, and training over the years. An objective measure of spasticity is required, and the development of robot-based systems for this purpose can help clinicians objectify their assessment.

It has been widely shown that robotic systems can be useful in the rehabilitation of adults and children with brain damage. In addition, these systems can be used to assess upper extremity function during treatment.

The aim in this study is to evaluate spasticity and hand grip strength with a finger hand robot in the Turkish population.

ELIGIBILITY:
Inclusion Criteria:

* Hemiplegic patients with sufficient cognitive and language skills to follow instructions will be included in the study.

Exclusion Criteria:

* Uncooperative Patient
* Having a skin ulcer on the hand,
* Patients with contractures of the hand fingers will be excluded.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 250 hemiplegia patients and 50 healthy controls aged between 40-85 years who applied to our clinic will be included in the study.
Sampling Method: Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Neurophysiological Evaluation | 2022.12-2023.1
  Brunnstrom Staging is a test that evaluates the motor development of hemiplegic patients. In this test, the neurophysiological recovery process of the hemiplegic patient was defined as 6 stages. According to this staging, the lowest stage; stage 1 (flask, the stage without voluntary movement), the highest stage was determined as stage 6 (stage with isolated joint movement). In Brunnstrom staging, the hand, upper extremity, and lower extremity are evaluated separately.
Muscle Power Assessment (MRC Scale) | 2022.12-2023.1
  The MRC is a scale for muscle strength that ranges from 0 to 5, relative to the maximum expected for a given muscle.
Spasticity Evaluation | 2022.12-2023.1
  It was planned to evaluate spasticity with the Modified Ashworth Scale (MAS). In MAS, patients are evaluated over 4 points. 0; there is no increase in muscle tone, and 4 indicates that the extremity is rigid in flexion and extension.
The Fugl-Meyer Assessment for Upper Extremity (FMA-UE) | 2022.12-2023.1
  The Fugl-Meyer Assessment Scale was developed to quantitatively evaluate sensorimotor recovery after stroke. It is based on Brunnstrom motor recovery stages. Turkish validity and reliability study was conducted.
Hand and Finger Grip Strength Assessment | 2022.12-2023.1
  Grip strength will be evaluated with the Jamar hydraulic hand dynamometer. Patients will be asked to squeeze with maximum force and each measurement will be made three times, and their averages will be recorded in kg. Finger grip strength will be evaluated with the "Jamar Digital Pinchmeter". Patients will be placed in the sitting position with the wrist in 90° flexion and the forearm in the neutral position. Measurements will be made bilaterally in three different positions as lateral, palmar and fingertip grips. Patients will be asked to squeeze with maximum force and each measurement will be made three times, and their averages will be recorded in kg. The dynamometer has a dual scale readout which displays isometric grip force from 0-90 kg. Higher scores means better grip strength.
Assessment with Amadeo Device | 2022.12-2023.1
  Amadeo (Tyromotion, Graz, Austria) is an end-effector device designed for the hand and is one of the very few options currently available on the commercial market. It is a device that is attached to the forearm with its groove-shaped structure and to the fingers with the support of magnets using bandages. The device performs flexion and extension movements of the fingers. It moves the fingers of the patients in the patterns defined in the software of the device. It provides training with passive, assistive and active movements that are ideal for use in all phases of neurological rehabilitation. It was planned to measure finger ROM, muscle strength and spasticity with Amadeo device.

CONTACTS AND LOCATIONS:
Overall Officials: Sevda ADAR, MD, Principal Investigator — Afyonkarahisar Health Sciences University; Ali İzzet AKÇİN, MD, Principal Investigator — Afyonkarahisar Health Sciences University
Locations (1):
- Afyonkarahisar Health Sciences University, Afyonkarahisar, Turkey (Türkiye)

REFERENCES:
- [Background] de-la-Torre R, Ona ED, Balaguer C, Jardon A. Robot-Aided Systems for Improving the Assessment of Upper Limb Spasticity: A Systematic Review. Sensors (Basel). 2020 Sep 14;20(18):5251. doi: 10.3390/s20185251. PMID 32937973
- [Background] Dehem S, Gilliaux M, Lejeune T, Detrembleur C, Galinski D, Sapin J, Vanderwegen M, Stoquart G. Assessment of upper limb spasticity in stroke patients using the robotic device REAplan. J Rehabil Med. 2017 Jul 7;49(7):565-571. doi: 10.2340/16501977-2248. PMID 28664214
- [Background] Luo Z, Lo WLA, Bian R, Wong S, Li L. Advanced quantitative estimation methods for spasticity: a literature review. J Int Med Res. 2020 Mar;48(3):300060519888425. doi: 10.1177/0300060519888425. Epub 2019 Dec 4. PMID 31801402